CLINICAL TRIAL: NCT01609790
Title: Phase II Double-Blinded Placebo-Controlled Study of Bevacizumab With or Without AMG 386 in Patients With Recurrent Glioblastoma or Gliosarcoma
Brief Title: Bevacizumab With or Without Trebananib in Treating Patients With Recurrent Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-01969; NCI-2012-01969 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S13-00759; CDR0000734205; RTOG-1122; RTOG-1122 (Other: NRG Oncology); RTOG-1122 (Other: CTEP); U10CA180868 (NIH); U10CA021661 (NIH)
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-05

CONDITIONS: Giant Cell Glioblastoma; Glioblastoma; Gliosarcoma; Oligodendroglioma; Recurrent Brain Neoplasm; Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Oligodendroglioma; Brain Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; trebananib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (bevacizumab and trebananib) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and trebananib IV over 30-60 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Biological: Trebananib
- Arm II (bevacizumab and placebo) (Active Comparator): Patients receive bevacizumab as in Arm I and placebo IV over 30-60 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may cross over to Arm I.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Placebo Administration

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; MYL-1402O; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Zirabev
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Placebo Administration — Given IV
  Arms: Arm II (bevacizumab and placebo)
Biological: Trebananib — Given IV
  Other Names: AMG 386; AMG386; Angiopoietin 1/2-Neutralizing Peptibody AMG 386
  Arms: Arm I (bevacizumab and trebananib)

SUMMARY:
This partially randomized phase II trial with a safety run-in component studies the side effects and how well bevacizumab given with or without trebananib works in treating patients with brain tumors that have come back (recurrent). Immunotherapy with monoclonal antibodies, such as bevacizumab, may induce changes in the body's immune system and interfere with the ability of tumor cells to grow and spread. Trebananib may stop the growth of tumor cells by blocking blood flow to the tumor. It is not yet known whether giving bevacizumab together with trebananib is more effective than bevacizumab alone in treating brain tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of AMG 386 (trebananib) 15 mg/kg weekly in combination with bevacizumab 10 mg/kg every 2 weeks (Cohort 1). (closed to accrual 10/2/12) II. To assess the efficacy of AMG 386 in combination with bevacizumab 10 mg/kg every 2 weeks compared to bevacizumab monotherapy in bevacizumab-naive patients, as measured by 6-month progression-free survival (PFS6) (Cohort 2).

SECONDARY OBJECTIVES:

I. To further assess the toxicity profile (Cohorts 1 and 2). II. To assess feasibility of AMG 386 15 mg/kg weekly in combination with bevacizumab 10 mg/kg every 2 weeks (Cohort 1 [closed to accrual 10/2/12]), as measured by the percentage of patients requiring dose reduction/interruption or discontinuation in the first 2 and subsequent cycles.

III. To determine the radiographic response rate (RR), median progression-free survival (PFS), and overall survival (OS) in bevacizumab-naive patients (Cohort 2).

IV. To assess the efficacy of AMG 386 15 mg/kg weekly in combination with bevacizumab 10 mg/kg every 2 weeks in patients who have progressed while on bevacizumab, as measured by overall survival (OS) (cross-over from placebo arm of Cohort 2).

V. To correlate outcome to treatment with tumor genotype, expression profile, and circulating angiogenesis biomarkers in tumor specimens (Cohort 2).

VI. To determine the RR, PFS6, and PFS in patients who have progressed while on bevacizumab therapy and receive AMG 386 in combination with bevacizumab (cross-over from placebo arm of Cohort 2).

VII. To determine the serum pharmacokinetics of AMG 386 in patients receiving bevacizumab (Cohort 1 and cross-over from placebo arm of Cohort 2).

OUTLINE: This is a safety study (cohort 1 [closed to accrual 10/2/12]) followed by a randomized study (cohort 2).

Cohort 1: Patients receive bevacizumab intravenously (IV) over 30-90 minutes on days 1 and 15 and trebananib IV over 30-60 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. (closed to accrual 10/2/12)

Cohort 2: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive bevacizumab and trebananib as in Cohort 1.

ARM II: Patients receive bevacizumab as in Arm I and placebo IV over 30-60 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may cross over to Arm I.

After completion of study treatment, patients are followed up at 30 days, every 2 months for 1 year, every 6 months for 1 year, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of glioblastoma or variants (gliosarcoma, glioblastoma with oligodendroglial features, giant cell glioblastoma); patients will be eligible if the original histology was a lower grade glioma and a subsequent histological diagnosis of glioblastoma or variants is made
* The tumor must be supratentorial; patients with infratentorial disease, spinal cord disease, and/or leptomeningeal disease are excluded
* Patients must have shown unequivocal evidence for tumor progression on the previous treatment regimen (prior to enrollment on this study) by magnetic resonance imaging (MRI) scan of the brain with and without contrast within 14 days prior to registration; the dose of steroids must be stable or decreasing for at least 5 days prior to the scan; patients with tumor progression who then undergo surgical resection prior to enrollment on study may be eligible as long as pathology confirms progressive or recurrent glioblastoma multiforme (GBM) (or variants); for patients who undergo surgical resection, registration on study may not occur any sooner than 28 days from surgery; an MRI scan of the brain with and without contrast is still required within 14 days prior to registration on study but is not required to demonstrate measurable disease or tumor progression after surgery
* Patients unable to undergo MRI because of non-compatible devices can be enrolled, provided computed tomography (CT) scans are obtained and are of sufficient quality; patients without non-compatible devices may not have CT scans performed to meet this requirement
* History/physical examination within 14 days prior to registration
* Karnofsky performance scale >= 70 within 14 days prior to registration
* Patients who have received prior treatment with interstitial brachytherapy, stereotactic radiosurgery, or implanted chemotherapy sources, such as wafers of polifeprosan 20 with carmustine, must have confirmation of progressive disease within 14 days prior to registration based upon nuclear imaging, magnetic resonance (MR) spectroscopy, perfusion imaging, or histopathology
* Leukocytes > 3,000/mm^3 (within 14 days prior to registration)
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3 (within 14 days prior to registration)
* Hemoglobin >= 10.0 g/dL (note: the use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 10.0 g/dL is acceptable) (within 14 days prior to registration)
* Platelets >= 100,000 cells/mm^3 (within 14 days prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 X institutional upper limit of normal (within 14 days prior to registration)
* Bilirubin =< 2.0 mg/dL (within 14 days prior to registration)
* Creatinine within normal upper institutional limits or creatinine clearance > 60 mL/min/1.73 m^2 (per 24 hour urine collection or calculated according to the Cockcroft-Gault formula) for subjects with creatinine levels above the institutional normal (within 14 days prior to registration)

  * Patients with creatinine levels below normal institutional limits are eligible
* Prothrombin time (PT)/international normalized ratio (INR) =< 1.5 (within 14 days prior to registration)
* Urinary protein =< 30 mg/dL in urinalysis or =< 1+ on dipstick (within 14 days prior to registration)
* Generally well-controlled blood pressure with systolic blood pressure =< 140 mm Hg AND diastolic blood pressure =< 90 mm Hg within 5 days prior to registration; the use of anti-hypertensive medications to control hypertension is permitted
* Women of childbearing potential must have a negative serum beta-human chorionic gonadotropin (HCG) pregnancy test within 14 days prior to registration
* Women of childbearing potential and male patients who are sexually active must practice adequate contraception during therapy and for 180 days (6 months) afterwards
* Patient must provide study specific informed consent prior to study entry

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible)
* Prior systemic cytotoxic chemotherapy within (i.e., =<) 28 days (42 days for nitrosoureas or mitomycin C) prior to registration, or patients who have not returned to baseline or =< Common Terminology Criteria for Adverse Events (CTCAE) version 4 (v. 4) grade 2 from adverse events (excluding alopecia) due to agents administered more than 28 days prior to registration
* Patients who received non-cytotoxic drug therapy must be off treatment for at least 14 days prior to registration; prior treatment with anti-vascular endothelial growth factor (VEGF) targeted agents; AMG 386 therapy; or other molecules that inhibit angiopoietins or TEK tyrosine kinase, endothelial (Tie2) receptor including, but not limited to, XL-820, XL-184 (cabozantinib-s-malate), and CVX-060/PF-4856884 is not allowed regardless of time frame
* Patients who have not yet completed at least 21 days (30 days for prior monoclonal antibody therapy) since ending other investigational device or drug trials, or who are currently receiving other investigational treatments
* Treatment within 30 days prior to enrollment with strong immune modulators, including but not limited to systemic cyclosporine, tacrolimus, sirolimus, mycophenolate mofetil, methotrexate, azathioprine, rapamycin, thalidomide, lenalidomide, and targeted immune modulators such as abatacept (CTLA-4-Ig), adalimumab, alefacept, anakinra, belatacept (LEA29Y), efalizumab, etanercept, infliximab, or rituximab
* Prior radiotherapy within 90 days (3 months) prior to registration unless there is either: a) histopathologic confirmation of recurrent tumor; or b) new enhancement on MRI outside of the radiation treatment field
* Major surgical procedure (including craniotomy and open brain biopsy) or significant traumatic injury within 28 days prior to registration or those patients who receive a non-central nervous system (CNS) minor surgical procedures (e.g. core biopsy or fine needle aspiration) within 3 days prior to registration; there is no waiting period for central line placement; there is a 7-day window for recovery prior to registration for patients who underwent stereotactic biopsy of the brain
* Prior therapy with anti-VEGF targeted agents (e.g. bevacizumab, cediranib, vandetanib, aflibercept, sunitinib, sorafenib, etc.); prior therapy with thalidomide and lenalidomide is allowed as long as treatment has not occurred within 30 days prior to enrollment
* More than 2 relapses
* Therapeutic anticoagulation with warfarin < 7 days prior to registration; (therapeutic or prophylactic therapy with aspirin, a low-molecular weight heparin, or a Factor Xa inhibitor is acceptable)
* Intratumoral hemorrhage or peritumoral hemorrhage, demonstrated by MRI or CT scan, CTCAE, v. 4 grade 2 or greater or evidence of significant hemorrhage (regardless of CTCAE, v. 4 grade) defined as > 1 cm diameter of blood (including postoperative hemorrhage)
* Gastrointestinal bleeding or any other hemorrhage/bleeding event CTCAE, v. 4 grade 3 or greater within 30 days prior to study entry
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within 180 days (6 months) prior to registration
  * Transmural myocardial infarction within 180 days (6 months) prior to registration
  * History of stroke, cerebral vascular accident (CVA), or transient ischemic attack within 180 days (6 months) prior to registration
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  * Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that human immunodeficiency virus (HIV) testing is not required for entry into this protocol
  * Known coagulopathy that increases risk of bleeding or a history of clinically significant hemorrhages in the past
  * History of non-healing wounds or ulcers, or bone fractures within 90 days (3 months) prior to registration
  * History of venous or arterial thromboembolism within 12 months prior to registration
* Prior allergic reaction to the study drugs involved in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2012-06-04 (Actual); Primary Completion 2015-10-02 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eudocia Q Lee, Principal Investigator — NRG Oncology
Locations (244):
- United States (243):
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Arizona Oncology-Deer Valley Center, Phoenix, Arizona
  - Arizona Oncology Services Foundation, Scottsdale, Arizona
  - Arizona Oncology Associates-West Orange Grove, Tucson, Arizona
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Sutter Cancer Research Consortium, Novato, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - William Backus Hospital, Norwich, Connecticut
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - New York Oncology Hematology PC - Albany, Albany, New York
  - New York Oncology Hematology PC - Albany Medical Center, Albany, New York
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Hematology Oncology Associates of Central New York-Liverpool, Liverpool, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Hematology Oncology Associates of Central New York-Rome, Rome, New York
  - Hematology Oncology Associates of Central New York-Onondaga Hill, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - Mountain Radiation Oncology PA, Asheville, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Messino Cancer Centers, Asheville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Warren Clinic Oncology-Tulsa, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Cancer Center-Natrona Heights, Natrona Heights, Pennsylvania
  - UPMC Jameson, New Castle, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Texas Oncology - South Austin Cancer Center, Austin, Texas
  - Texas Oncology Bedford, Bedford, Texas
  - Texas Oncology at Baylor Charles A Sammons Cancer Center, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - Texas Oncology-Grapevine, Grapevine, Texas
  - Texas Oncology-Longview Cancer Center, Longview, Texas
  - Texas Oncology-Seton Williamson, Round Rock, Texas
  - Texas Oncology - Round Rock Cancer Center, Round Rock, Texas
  - Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Tyler Cancer Center, Tyler, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Cancer Care Northwest-North Spokane, Spokane, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada

REFERENCES:
- [Derived] Lee EQ, Zhang P, Wen PY, Gerstner ER, Reardon DA, Aldape KD, deGroot JF, Pan E, Raizer JJ, Kim LJ, Chmura SJ, Robins HI, Connelly JM, Battiste JD, Villano JL, Wagle N, Merrell RT, Wendland MM, Mehta MP. NRG/RTOG 1122: A phase 2, double-blinded, placebo-controlled study of bevacizumab with and without trebananib in patients with recurrent glioblastoma or gliosarcoma. Cancer. 2020 Jun 15;126(12):2821-2828. doi: 10.1002/cncr.32811. Epub 2020 Mar 10. PMID 32154928

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Safety Run-In; Cohort 2: Bevacizumab+AMG 386: Bevacizumab every 2 weeks + AMG 386 weekly until disease progression.
- Cohort 2: Bevacizumab+Placebo: Bevacizumab every 2 weeks + placebo weekly until disease progression. Patients who progress will be allowed to cross over and receive treatment with bevacizumab + AMG 386
Period: Overall Study
Arm/Group | Cohort 1: Safety Run-In | Cohort 2: Bevacizumab+Placebo | Cohort 2: Bevacizumab+AMG 386
Started | 7 | 65 | 65
Completed | 6 (Subjects with data available for analysis are considered to have completed the study.) | 58 (Subjects with data available for analysis are considered to have completed the study.) | 57 (Subjects with data available for analysis are considered to have completed the study.)
Not Completed | 1 | 7 | 8
Not completed — Protocol Violation | 1 | 7 | 8

BASELINE CHARACTERISTICS:
Population: All eligible patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Safety Run-In | Cohort 2: Bevacizumab+Placebo | Cohort 2: Bevacizumab+AMG 386 | Total
Number analyzed (Participants) | 6 | 58 | 57 | 121
Age, Continuous [Median (Full Range); unit: years] | 56 [28 to 75] | 58 [22 to 79] | 57 [30 to 80] | 58 [22 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 22 | 25 | 48
  Male | 5 | 36 | 32 | 73

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing of Dose-limiting Toxicity (Cohort 1)
Description: Dose-limiting toxicity (DLT), defined as a clinically significant adverse event or abnormal laboratory value assessed as unrelated to disease progression, intercurrent illness, or concomitant medications and meets any of the criteria below. Any DLT must be a toxicity possibly related to protocol treatment during first 4 weeks: grade 4 hematologic toxicity, grade 3/4 thrombocytopenia, or grade 3/4 non-hematologic toxicity; Gastrointestinal fistula, bowel perforation, intracranial hemorrhage, wound dehiscence, or reversible posterior leukoencephalopathy of any grade; Delay of treatment > 28 days. If 2+ of patients experience a DLT among 6 eligible patients, this drug combination will be considered unsafe and a lower dose of AMG will be explored; otherwise conclude that this drug combination is safe. The probability of claiming safe dose is no more than 16% when the true DLT rate is >45%, and the probability of claiming safe dose is at least 78% when the true DLT rate is <= 15%.
Time Frame: From start of treatment to 4 weeks.
Population: All eligible patients who started study treatment
Measure: Number; unit: participants
Groups:
- Safety Run-In: Bevacizumab every 2 weeks + AMG 386 weekly until disease progression.
Arm/Group | Safety Run-In
Number analyzed (Participants) | 6
participants | 0

2. Primary Outcome: Six-month Progression-free Survival (Cohort 2)
Description: As determined by central review of MRI exams, assessed using RANO criteria for progression that is defined by any of the following: > 25% increase in sum of the products of perpendicular diameters of enhancing lesions compared to the smallest tumor measurement obtained either at baseline (if no decrease) or best response, on stable or increasing doses of corticosteroids; Significant increase in T2/FLAIR non-enhancing lesion on stable or increasing doses of corticosteroids compared to baseline scan or best response following initiation of therapy, not due to co-morbid events; Any new lesion; Clear clinical deterioration not attributable to other causes apart from the tumor or changes in corticosteroid dose; Failure to return for evaluation due to death or deteriorating condition; Clear progression of non-measurable disease.
Time Frame: From randomization to six months.
Population: Randomized patients evaluable for 6 months progression-free survival (PFS).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: Bevacizumab+Placebo | Cohort 2: Bevacizumab+AMG 386
Number analyzed (Participants) | 56 | 53
percentage of participants | 41.1 [28.2 to 54.0] | 22.6 [11.4 to 33.9]
Statistical Analysis 1: Comparison: Cohort 2: Bevacizumab+Placebo vs Cohort 2: Bevacizumab+AMG 386; Assuming a 36% 6-month (6m) rate in the placebo arm [from the March 2009 Food and Drug Administration (FDA) briefing], a 55% rate in the AMG 386 arm, and an exponential distribution corresponds to median PFS of 4.1 and 7 months, respectively, with a hazard ratio of 0.59 (AMG 386 arm vs. placebo arm). A total of 114 patients (57 per arm) will yield 85% power to detect an absolute 19% difference of 6m PFS rate at a 1-sided alpha level of 0.15 based on a 2-sample proportion test; Test type: Superiority or Other; p = 0.98, Z-test; One-sided test, significance level 0.15

3. Secondary Outcome: Incidence of Grade 3+ Treatment-related Toxicity, Measured by CTCAE v. 4 (Cohort 2)
Description: Adverse events (AEs) are graded by using CTCAE 4.0. Possibly/probably/definitely related to protocol treatment AEs are considered.
Time Frame: From start of treatment up to 3 years.
Population: Randomized and eligible patients who started protocol treatment.
Measure: Number; unit: participants
Arm/Group | Cohort 2: Bevacizumab+Placebo | Cohort 2: Bevacizumab+AMG 386
Number analyzed (Participants) | 57 | 57
participants | 21 | 20
Statistical Analysis 1: Comparison: Cohort 2: Bevacizumab+Placebo vs Cohort 2: Bevacizumab+AMG 386; Test type: Superiority or Other; p = 0.85, Chi-squared

4. Secondary Outcome: Overall Survival (Cohort 2)
Description: Survival time is defined as time from randomization to date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact. This analysis was planned to occur when all patients had been potentially followed for at least 6 months.
Time Frame: From randomization up to 3 years.
Population: All randomized and eligible patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 2: Bevacizumab+Placebo | Cohort 2: Bevacizumab+AMG 386
Number analyzed (Participants) | 58 | 57
Months | 11.5 [8.4 to 14.2] | 7.5 [6.8 to 10.1]
Statistical Analysis 1: Comparison: Cohort 2: Bevacizumab+Placebo vs Cohort 2: Bevacizumab+AMG 386; Test type: Superiority or Other; p = 0.09, Log Rank; Hazard Ratio (HR) = 1.46, 95% CI 2-sided [0.95 to 2.27]

5. Secondary Outcome: Progression-free Survival (Cohort 2)
Description: Progression-free survival time is measured from randomization to the date of first progression or death or, otherwise, the last follow-up date on which the patient was reported alive. This analysis was planned to occur when all patients had been potentially followed for at least 6 months.
Time Frame: From randomization up to 3 years.
Population: All randomized and eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: Bevacizumab+Placebo | Cohort 2: Bevacizumab+AMG 386
Number analyzed (Participants) | 58 | 57
percentage of participants | 4.8 [3.8 to 7.1] | 4.2 [3.7 to 5.6]
Statistical Analysis 1: Comparison: Cohort 2: Bevacizumab+Placebo vs Cohort 2: Bevacizumab+AMG 386; Test type: Superiority or Other; p = 0.04, Log Rank; Hazard Ratio (HR) = 1.51, 95% CI 2-sided [1.02 to 2.24]

6. Secondary Outcome: Radiographic Response Rate (Cohort 2)
Description: Proportion of patients with best overall response of complete response (CR) or partial response (PR) recorded from the start of the treatment until disease progression/recurrence. Response determined by site-reported radiology review of MRI exams using Response Assessment in Neuro-Oncology Criteria (RANO) criteria. CR: Complete disappearance of all enhancing measurable disease (MD) + non-measurable disease (NMD) sustained >= 4 wks; No new lesions; Stable or improved non-enhancing (T2/FLAIR) lesions; Off corticosteroids (or on physiologic replacement doses only); Stable/improved clinically. PR: >= 50% decrease vs. baseline of sum of products of perpendicular diameters of all measurable enhancing lesions sustained >= 4 wks; No progression of NMD; No new lesions; Stable/improved non-enhancing (T2/FLAIR) lesions on <= dose of corticosteroids vs. baseline scan; Corticosteroid dose at evaluation scan <= baseline scan dose; Stable or improved clinically. NMD only cannot be a CR or PR.
Time Frame: From randomization up to 3 years.
Population: All randomized and eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: Bevacizumab+Placebo | Cohort 2: Bevacizumab+AMG 386
Number analyzed (Participants) | 58 | 57
percentage of participants | 5.9 [0 to 12.3] | 4.2 [0 to 9.8]
Statistical Analysis 1: Comparison: Cohort 2: Bevacizumab+Placebo vs Cohort 2: Bevacizumab+AMG 386; Test type: Superiority or Other; p = 0.7, Chi-squared

7. Secondary Outcome: Percentage of Patients Requiring Dose Reduction/Interruption or Discontinuation in the First 2 and Subsequent Courses (Cohort 1)
Description: Feasibility of trebananib weekly in combination with bevacizumab every 2 weeks, measured by the percentage of patients requiring dose reduction/interruption or discontinuation in the first 2 and subsequent courses (Cohort 1)
Time Frame: From randomization up to 3 years.
Population: Eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Run-In
Number analyzed (Participants) | 6
Participants
  In first 2 cycles | 6
  In first 6 cycles | 3
  In first 12 cycles | 5

8. Other Pre Specified Outcome: Tumor Genotype, Expression Profile, and Circulating Angiogenesis Biomarkers (Cohort 2)
Description: Biomarker data has not yet been obtained and therefore this outcome measure cannot yet be reported.
Time Frame: From randomization to date of death or last followup. Statistical analysis occurs when tumor genotype, expression profile and circulating angiogenesis biomarkers have been determined from the tissue specimens.
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Randomized and eligible patients who started protocol treatment are included in the adverse event tables. Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | Cohort 1: Safety Run-In | Cohort 2: Bevacizumab+Placebo | Cohort 2: Bevacizumab+AMG 386
Serious Adverse Events (participants affected / at risk) | 5/6 | 22/57 | 20/57
Other Adverse Events (participants affected / at risk) | 6/6 | 57/57 | 54/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Safety Run-In (N=6) | Cohort 2: Bevacizumab+Placebo (N=57) | Cohort 2: Bevacizumab+AMG 386 (N=57)
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Edema limbs (General disorders) | 0 | 1 | 1
Flu like symptoms (General disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 3 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Infections and infestations - Other (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 1 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 3 | 0
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 3
Aphonia (Nervous system disorders) | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 1 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 2 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 2 | 0
Encephalopathy (Nervous system disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 1 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 1 | 1
Memory impairment (Nervous system disorders) | 0 | 1 | 0
Nervous system disorders - Other (Nervous system disorders) | 0 | 0 | 2
Seizure (Nervous system disorders) | 2 | 4 | 4
Stroke (Nervous system disorders) | 0 | 2 | 1
Transient ischemic attacks (Nervous system disorders) | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 2 | 3
Delirium (Psychiatric disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 3
Thromboembolic event (Vascular disorders) | 0 | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Safety Run-In (N=6) | Cohort 2: Bevacizumab+Placebo (N=57) | Cohort 2: Bevacizumab+AMG 386 (N=57)
Anemia (Blood and lymphatic system disorders) | 3 | 14 | 9
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 2
Cushingoid (Endocrine disorders) | 1 | 0 | 2
Blurred vision (Eye disorders) | 0 | 4 | 7
Dry eye (Eye disorders) | 1 | 1 | 1
Eye disorders - Other (Eye disorders) | 0 | 5 | 9
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 5
Constipation (Gastrointestinal disorders) | 3 | 15 | 6
Diarrhea (Gastrointestinal disorders) | 2 | 13 | 8
Dry mouth (Gastrointestinal disorders) | 0 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 6 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 3
Fecal incontinence (Gastrointestinal disorders) | 1 | 2 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 3 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 4 | 4
Nausea (Gastrointestinal disorders) | 2 | 14 | 8
Vomiting (Gastrointestinal disorders) | 2 | 11 | 2
Chills (General disorders) | 0 | 3 | 0
Edema face (General disorders) | 0 | 1 | 4
Edema limbs (General disorders) | 2 | 12 | 12
Fatigue (General disorders) | 4 | 38 | 37
Fever (General disorders) | 1 | 6 | 0
Gait disturbance (General disorders) | 1 | 13 | 7
General disorders and administration site conditions - Other (General disorders) | 0 | 4 | 2
Injection site reaction (General disorders) | 1 | 1 | 1
Localized edema (General disorders) | 0 | 4 | 1
Malaise (General disorders) | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 2 | 2
Pain (General disorders) | 2 | 8 | 8
Esophageal infection (Infections and infestations) | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 3 | 3
Urinary tract infection (Infections and infestations) | 1 | 1 | 4
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 4 | 4
Fall (Injury, poisoning and procedural complications) | 2 | 5 | 9
Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 2 | 3
Alanine aminotransferase increased (Investigations) | 3 | 15 | 9
Alkaline phosphatase increased (Investigations) | 2 | 5 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 9 | 6
Blood bilirubin increased (Investigations) | 0 | 3 | 3
CPK increased (Investigations) | 1 | 0 | 0
Creatinine increased (Investigations) | 1 | 1 | 2
Investigations - Other (Investigations) | 1 | 3 | 3
Lymphocyte count decreased (Investigations) | 2 | 17 | 15
Neutrophil count decreased (Investigations) | 0 | 6 | 4
Platelet count decreased (Investigations) | 1 | 10 | 10
Weight gain (Investigations) | 1 | 0 | 3
Weight loss (Investigations) | 2 | 6 | 2
White blood cell decreased (Investigations) | 1 | 11 | 10
Anorexia (Metabolism and nutrition disorders) | 2 | 10 | 5
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 22 | 16
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 4 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 3 | 5
Hypernatremia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 5 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 3 | 5
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 1 | 8 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 6 | 4
Hyponatremia (Metabolism and nutrition disorders) | 2 | 9 | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 8 | 5
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 11 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 7 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 9 | 10
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 12 | 6
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 5 | 8
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 3 | 4
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 9 | 9
Amnesia (Nervous system disorders) | 1 | 1 | 2
Ataxia (Nervous system disorders) | 2 | 5 | 4
Cognitive disturbance (Nervous system disorders) | 0 | 8 | 2
Concentration impairment (Nervous system disorders) | 1 | 0 | 2
Depressed level of consciousness (Nervous system disorders) | 1 | 2 | 0
Dizziness (Nervous system disorders) | 2 | 11 | 11
Dysarthria (Nervous system disorders) | 0 | 6 | 6
Dysgeusia (Nervous system disorders) | 1 | 0 | 1
Dysphasia (Nervous system disorders) | 1 | 10 | 7
Facial muscle weakness (Nervous system disorders) | 2 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 32 | 19
Lethargy (Nervous system disorders) | 1 | 1 | 1
Memory impairment (Nervous system disorders) | 1 | 11 | 10
Nervous system disorders - Other (Nervous system disorders) | 1 | 9 | 7
Paresthesia (Nervous system disorders) | 1 | 7 | 8
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 5 | 5
Seizure (Nervous system disorders) | 1 | 11 | 5
Somnolence (Nervous system disorders) | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 5 | 3
Agitation (Psychiatric disorders) | 1 | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 9 | 4
Confusion (Psychiatric disorders) | 3 | 7 | 6
Depression (Psychiatric disorders) | 1 | 9 | 9
Insomnia (Psychiatric disorders) | 3 | 9 | 11
Hematuria (Renal and urinary disorders) | 2 | 5 | 5
Proteinuria (Renal and urinary disorders) | 1 | 9 | 7
Urinary frequency (Renal and urinary disorders) | 2 | 3 | 4
Urinary incontinence (Renal and urinary disorders) | 3 | 5 | 4
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 12 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 7 | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 4
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 3 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 6
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 4
Purpura (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 4 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 5 | 2
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 5 | 3
Hematoma (Vascular disorders) | 2 | 1 | 1
Hypertension (Vascular disorders) | 3 | 24 | 25
Thromboembolic event (Vascular disorders) | 1 | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less